CLINICAL TRIAL: NCT07342387
Title: Development of Microfluidic Patch-type Sweat Sensor Utilizing Surface-enhanced Raman Mechanism
Brief Title: Development of Microfluidic Patch-type Sweat Sensor
Acronym: sweat sensor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Korea University (Other)
Responsible Party: Principal Investigator, LEE SUNGHO, Professor, Korea University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2024AN0368
Record Dates: First submitted 2026-01-08; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Diseases of the Genitourinary System
MeSH Terms: conditions — Urogenital Diseases | interventions — Sodium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group (Experimental): Measurement of creatinine concentration in sweat using a microfluidic patch-based sweat sensor
  Interventions: Other: Time-course changes in Sodium and Creatinine levels.

INTERVENTIONS:
Other: Time-course changes in Sodium and Creatinine levels. — Time-course changes in Sodium and Creatinine levels.

SUMMARY:
1. Background Value of Sweat: Sweat has gained significant attention as a key biomarker for diagnosing dehydration and renal dysfunction (e.g., uremia), as it contains essential indicators that reflect blood concentrations, such as electrolytes and metabolites (creatinine, urea).

Technical Transition: To overcome the limitations of conventional absorbent pads, such as contamination and evaporation, it is essential to develop flexible, wearable microfluidic devices that enable immediate collection and high-precision analysis.

Domestic and International Trends: While countries like the U.S. are already utilizing real-time IoT monitoring technologies in military and sports sectors, there is an urgent need in Korea to secure physiological data optimized for the Korean population and to establish a robust medical analysis system.

2. Objectives To develop a skin-interfaced microfluidic platform integrated with a SERS biosensor for high-sensitivity, real-time detection of Sodium and Creatinine to monitor dehydration and renal health.

3. Research Plan

1. Subject Selection: Recruit and obtain informed consent from patients visiting the hospital with renal disease (creatinine levels 1.5 mg/dL or higher).
2. Clinical Schedule: Conduct the clinical study on the subjects' scheduled routine blood test dates.
3. Patch Attachment: Apply the sweat collection patch and a control absorption pad to 1-2 body areas (e.g., center of the chest, forehead).
4. Sweat Induction: Induce sweating by having subjects wait in an electric thermal chamber for 30 minutes.
5. Absorption Pad Collection: For the control pads (which cannot collect time-series data), attach two initially and retrieve them during the early stages of sweat secretion.
6. Microfluidic Patch Collection: Measure the volume of sweat collected (~100 uL per subject) to calculate sweat loss, then seal and transport to the laboratory.
7. Comparative Sample Processing: Measure the weight of absorption pads before/after use to determine fluid loss. Extract sweat samples (~500 uL per subject) into micro-tubes for transport.
8. Contamination Control: Utilize dry ice and insulated coolers during transport to prevent sample degradation or contamination.
9. Quantitative Analysis & Evaluation: Perform quantitative analysis of sodium and creatinine levels from both samples using the proposed SERS-based method and standard analytical tools (HPLC or LC-MS). Compare the changes in biomarkers and sweat loss over time to evaluate and summarize the hydration status and renal function patterns of each subject.

ELIGIBILITY:
Inclusion Criteria:

* Aged 19 years or older
* Patients with renal disease and a blood (serum) creatinine level of 1.5 mg/dL or higher

Exclusion Criteria:

* Subjects who do not provide consent to participate in this study
* Subjects with a medical history of skin allergies related to patches/adhesives

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2024-06-15 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2026-01-07 (Actual)

PRIMARY OUTCOMES:
Time-course changes in Sodium and Creatinine levels. | enrollment day
  Measurement on the day of enrollment (Visit 1), followed by study termination

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Anam Hospital, Seoul, Seongbuk-gu, South Korea

IPD SHARING:
Plan to Share IPD: No